CLINICAL TRIAL: NCT00534924
Title: The Effects of Post-Conditioning and Administration of Vitamin C on Intramuscular High Energy Phosphate Levels
Acronym: IRI in MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2007-002520-16
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Ischemia Reperfusion Injury
Keywords: IR injury; MRI; Vitamin C; Postconditioning
MeSH Terms: conditions — Reperfusion Injury | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): No intervention after IR injury
  Interventions: Other: no intervention
- 2 (Experimental): Postconditioning
  Interventions: Procedure: Postconditioning
- 3 (Experimental): Vit. C
  Interventions: Drug: Vit C

INTERVENTIONS:
Drug: Vit C
  Arms: 3
Procedure: Postconditioning
  Arms: 2
Other: no intervention
  Arms: 1

SUMMARY:
Ischemic injury to muscular tissue is common in cardiovascular medicine. The most effective treatment to avoid ischemic damage is the rapid re-establishment of reperfusion. However, reperfusion itself can result in additional damage to ischemic tissue. This phenomenon is called ischemia - reperfusion (IR) injury and is caused by different pathologic mechanisms.

Therapies are required which can be administered after the onset of an ischemic event to protect the tissue against IR injury. Therefore, a promising strategy to reduce IR injury is post-conditioning.

Likewise, pharmacological therapies administered after the onset of reperfusion might prevent tissue injury. We have recently shown that high concentrations of exogenous vitamin C abrogate experimental IR injury of the forearm vasculature in patients with peripheral artery disease and in healthy subjects.

Study hypothesis

We hypothesize that the administration of mechanical post-conditioning or of high-dose vitamin C may protect skeletal muscle against IR injury. This shall be studied employing MR spectroscopy of the leg, which is an established model to assess muscle aerobic energy metabolism.

Design

Three periods, three way cross over study in 10 volunteers. One screening visit, three one-day study days with two washout periods of >3 days in between are scheduled for each participant. The order of experimental days will be randomized. After the last treatment a final follow-up examination will be performed within one week.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 45 years
* Nonsmoker for more than 3 months
* Body mass index between 18 and 25 kg/m2
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

Any of the following will exclude a subject from the study:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia
* Treatment in the previous 3 weeks with any drug including over-the-counter drugs.
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* History or presence of gastrointestinal, liver of kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of the study drug
* Blood donation during the previous 3 weeks
* History of hypersensitivity to parenteral vitamin C.
* Glucose-6-phosphate dehydrogenase deficiency
* Thalassemia, haemochromatosis
* History of urolithiasis
* Any metallic or paramagnetic device not removable
* Claustrophobia
* Regular use of supplementary oral Vitamin C or Vitamin C containing substances

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Prof., Principal Investigator — Head of research group
Locations (1):
- Medical University of Vienna, Vienna, Austria